CLINICAL TRIAL: NCT02996955
Title: Influence of Social Support and Treatment of Illness Perceptions on Patient's Adherence to a Physical Activity Advice
Brief Title: Patient Adherence to a Physical Activity Advice
Acronym: PAPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NL58005.096.16
Record Dates: First submitted 2016-11-29; First posted 2016-12-19 (Estimated); Last update posted 2024-04-19 (Actual); Status verified 2024-01

CONDITIONS: Patient Adherence
Keywords: Low Back Pain; Social Support; Illness Perceptions; Activity Advice
MeSH Terms: conditions — Patient Compliance; Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- SoSup group (Experimental): usual care will be provided and social support and treatment of illness perceptions and activity advice and wearing the activ8
  Interventions: Behavioral: social support; Behavioral: treatment of illness perceptions; Device: Activ8; Other: activity advice
- C group (Active Comparator): usual care will be provided and treatment of illness perceptions and activity advice and wearing the Activ8
  Interventions: Behavioral: treatment of illness perceptions; Device: Activ8; Other: activity advice

INTERVENTIONS:
Behavioral: social support — behaviour change intervention
  Arms: SoSup group
Behavioral: treatment of illness perceptions — educational interview
Device: Activ8 — wearing a move monitor
Other: activity advice — walking or cycling 5 days a week during at least half an hour

SUMMARY:
Low back pain is worldwide a common musculoskeletal condition with a high number of recurrences. Recurrence rate and the number of recurrences could be reduced and time to a next episode could be prolonged by advising an active lifestyle. Advising regular physical activity is the mainstay in physical therapy treatment. This includes an appeal to patients to adhere to an activity advice. Patient adherence to an activity advice is poor. In this study an intervention consisting of treatment of illness perceptions with or without organizing social support to increase adherence to an activity advice will be investigated.

The primary objective of this study is to investigate whether social support by a partner or friend and treatment of patients' illness perceptions influences the rate of adherence to an activity advice compared to treatment of patients' illness perceptions alone in patients suffering non-specific low back pain. Secondary objectives are; a) whether 'treatment of illness perceptions' changes patients' maladaptive illness perceptions into realistic ones, b) whether maladaptive illness perceptions, comorbidity and/or overweighed/obesity and/or rate of recurrences of non-specific low back pain and/or attitude and intention to physical activity influences patient's adherence .

This study is a multi-centre randomized two-arm controlled clinical trial. Patients ≥18 years presenting with at least a second episode of non-specific low back pain.

Patients in the intervention and control group will be asked to perform a physical activity advice. During two physiotherapy treatment sessions treatment of illness perceptions is performed in both groups. In the intervention group organizing social support by a partner or friend is added.

Twenty-five percent absolute improvement of walking and/or cycling according the NNGB in the intervention group is clinically relevant.

During four appointments several questionnaires have to be filled in and during two physiotherapy treatment sessions half an hour treatment of illness perceptions will be performed. Social support by a partner or friend will be organized during the same physiotherapy treatment sessions in the intervention group. During three separate weeks patients have to wear an activity monitor. Patients will be treated according to the Dutch Low Back Pain guideline; no adverse effects will be expected.

DETAILED DESCRIPTION:
Objective of the study:

The primary objective of this study is to investigate whether social support by a partner or friend and treatment of patients' illness perceptions influences the rate of adherence to an activity advice compared to treatment of patients' illness perceptions alone in patients suffering non-specific low back pain. Secondary objectives are; 1) Whether 'treatment of illness perceptions' changes patients' maladaptive illness perceptions into realistic ones, 2) Whether maladaptive illness perceptions, comorbidity and/or obesity and/or rate of recurrences of non-specific low back pain and/or attitude and intention to physical activity influences patient's adherence to an activity advice.

Study design:

This study is a multicentre randomized two arm, controlled clinical trial. During a twelve-week intervention period, one group of patients will receive an activity advice added to usual treatment including 'treatment of illness perceptions' (C-group). The other group will receive an activity advice and the intervention addressing social support by a partner or friend added to usual treatment including 'treatment of illness perceptions' (SoSup-group). Patients will be assessed at baseline, and after one, 6 and 12 weeks. Recruitment is scheduled from October 2016 to July 2017. The study will be performed in 12 centres for physiotherapy in the province Zuid-Holland, the Netherlands.

Study population:

It is mentioned that individuals with recurrent non-specific low back pain score more unfavourable on lifestyle risk factors including physical inactivity than individuals without or first time non-specific low back pain (van Oostrom et al., 2012). To include potential physically inactive non-specific low back pain sufferers, patients ≥18 years presenting with at least a second episode of non-specific low back pain who are not physical active in accordance with the NNGB are recruited for the study.

Intervention (if applicable):

In both the C- and SoSup-group an activity advice will be added to usual treatment. The advised activities will be walking and/or cycling outdoors, meeting the Dutch Standard Healthy Physical Activity (NNGB) (Hildebrandt et al., 2007). In both groups cognitive treatment on illness perceptions according to the common sense model to the patient in the presence of the partner or friend will be given. During a maximum of two half-hour contacts in a standardised dialogue on maladaptive beliefs and feelings about identity, time-line, causes, controllability, and curability of low back pain are mapped, maladaptive perceptions are challenged, alternative perceptions are formulated (Siemonsma et al., 2013). The intervention in the SoSup-group (intervention group), organizing social support by a partner or friend depending on patient's preferences, will be added. During a maximum of two half-hour contacts (one for explanation and one for evaluation), in a standardised discussion the partner or friend will be stimulated to support the patient in executing the activity advice. During 12 weeks the social support by a partner or friend will be executed for at least 5 times a week.

Primary study parameters/outcome of the study:

The primary outcome measure will be walking and/or cycling according to the NNGB and social support.

Secundary study parameters/outcome of the study (if applicable):

Other outcomes will be 1. measures of illness perceptions. 2. measures of comorbidity, BMI, number of recurrences of non-specific low back pain, measures of attitude and intention to physical activity 3. measures of refusal of the study.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness (if applicable):

The social support described in this study is designed for better outcomes of physical activity levels patients suffering low back pain, and has no proven advantage on better outcomes on pain and disability in non-specific low back pain sufferers. Therefore we consider there is no disadvantage in the SoSup-group versus the C-group because patients in both groups receive concomitant best evidence healthcare according to the Dutch guideline for low back pain (Staal et al., 2013). No adverse effects of the interventions are expected. There are no ethical implications to be expected as a result of this study, treatment of all patients during the intervention period will be according to the Dutch guideline for low back pain.

ELIGIBILITY:
Inclusion Criteria:

• Non-specific low back pain

Exclusion Criteria:

* Patients physical active in accordance with the Dutch Standard Healthy Physical Activity (NNGB) (Hildebrandt et al., 2007)
* Patients with specific low back pain
* Onset of the low back pain after age 50 years,
* Continuous pain regardless of posture or movement,
* Nocturnal pain,
* General malaise,
* History of malignancy,
* Unexplained weight loss,
* Elevated erythrocyte sedimentation rate (ESR)
* Previous vertebral fracture,
* Older person with hip fracture,
* Prolonged use of corticosteroids,
* Onset of low back pain before age 20 years,
* Iridocyclitis,
* History of unexplained peripheral arthritis or inflammatory bowel disease,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
adherence to the activity advice | 12 weeks
  proportion of patients (non)adhering to the activity advice measured by the Activ8

SECONDARY OUTCOMES:
changes in patient's illness perceptions | base line, one week, 6 and 12 weeks
  proportion of patients with (un)changed illness perceptions measured by the Brief Illness Perception Questionnaire- short, Dutch version.

OTHER OUTCOMES:
influence of illness perception on adherence | 12 weeks
  proportion of patients with (mal)adaptive illness perception measured by the BIPQ-s Dutch version (non)adhering the activity advice measured by the Activ8
influence of comorbidity on adherence | 12 weeks
  proportion of patients with or without comorbidity measured by the Cumulative Illness Rating Scale (non)adhering the activity advice measured by the Activ8
influence of overweight/obesity on adherence | 12 weeks
  proportion of patients with or without overweight/obesity measured with Body Mass Index (non)adhering the activity advice measured by the Activ8
influence of number of episodes of low back pain on adherence | 12 weeks
  proportion of patients with or without more than 2 episodes low back pain (non)adhering the activity advice measured by the activ8
change of influence of attitude and intention to a physical activity on adherence | base line, one week, 6 and 12 weeks
  proportion of patients with or without adequate atitude/intention to physical activity measured by the Module Houding en Intentie Questionnaire (non)adhering the activity advice measured by the activ8
influence of perceived pain and disability on adherence | base line
  proportion of patients with or without high scores on VAS pain and Quebec Back Pain and Disability scale (non) adhering the activity advice measured by the activ8

CONTACTS AND LOCATIONS:
Overall Officials: Rob de Bie, Prof. PhD, Study Chair — Maastricht University; Henk v Mameren, Em Prof PhD, Study Chair — Maastricht University
Locations (1):
- Maastricht University, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] van Koppen B, Zandwijk P, van Mameren H, de Bie R. Patient adherence to physical activity advice (PAPA) in patients with low back pain: Study protocol for a multicentre randomized controlled trial. Physiother Res Int. 2022 Oct;27(4):e1969. doi: 10.1002/pri.1969. Epub 2022 Aug 17. PMID 35975659